CLINICAL TRIAL: NCT01907035
Title: Improving Anxiety-depressive Disorder in Primary Care Applying a Cognitive-behavioral Treatment, Applied by Psychologists.
Brief Title: Anxiety-depressive Disorder in Primary Care and Cognitive-behavioral Treatment
Acronym: PSICCAPAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Amale Jauregui Larrabeiti, IPrincipal Investigator, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSICCAPAD 2012; 2011111064 (Other Grant/Funding Number: Basque Health departament)
Record Dates: First submitted 2013-07-22; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Anxiety-depressive Patients Mild to Moderate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-behavioral intervention (Experimental): Cognitive-behavioral intervention: Evaluate the effectiveness of a cognitive-behavioral intervention by psychologists in collaboration with practitioner plus routine therapy in the field of primary care in anxiety-depressive patients mild to moderate, with respect to standardized usual care by physicians, improve quality of life of these people, producing at least ten-point increase in the level of overall quality of life (SF-36)
  Interventions: Behavioral: A cognitive-behavioral intervention
- Usual care (Active Comparator): Family practice attention without the psychologist support
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: A cognitive-behavioral intervention — Evaluate the effectiveness of a cognitive-behavioral intervention by psychologists in collaboration with MF plus routine therapy in the field of APS in anxiety-depressive patients mild to moderate, with respect to standardized usual care by physicians, improve quality of life of these people, producing at least ten-point increase in the level of overall quality of life (SF-36)
  Arms: Cognitive-behavioral intervention
Other: Usual care
  Arms: Usual care

SUMMARY:
OBJECTIVE: Evaluate the effectiveness of quality of life score, a cognitive-behavioral intervention by psychologists in the field of primary care in anxiety-depressive patients, mild to moderate, compared with usual care.

DESIGN: Clinical trial, multicenter, prospective, and randomized into two parallel groups. SCOPE AND SUBJECTS: We included a random sample of 246 patients anxious-depressive, mild / moderate, belonging to the target population of 41 doctors from several health centers. INTERVENTION: In the 246 patients randomly assigned to the intervention group, with a standardized program of cognitive behavioral therapy applied by psychologists, by the usual treatment or control group, which will be standard care. MEASUREMENTS: The main result will be changes in general health scores of the SF-36. It will also measure the change in frequency and intensity of anxiety-depressive symptoms on the scales HARS, HDRS, STAI and BDI at baseline and at 2, 6 and 12 months. In addition, also collected for drug use and health services.

ANALYSIS: Analyses were performed by intention to treat, comparing the change obtained in both groups at the end of the 12 month follow up. Estimates of the effect attributable to the intervention by the difference in those changes, adjusting in addition to the baseline, the possible confounding covariates or effect modifiers of the intervention, using longitudinal mixed-effects models.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patients.
* Adults.
* Of both sexes.
* With disorder mixed anxiety-depressive mild-moderate active diagnosed by their general practitioner and showing more than 4 points in Goldberg-Anxiety, and more than 3 in Goldberg Depression.

Exclusion Criteria:

* Patients under 18 or over 75 years
* Patients with inability to understand, read or speak Spanish
* Patients with cognitive impairment
* Patients with severe disease which in the opinion of your doctor have a presumably fatal end during the 12 month follow-up
* Patients with psychotic disorders or other serious mental disease
* Patients with attempted suicide or suicidal ideation persistent
* Patients referred to Specialized Care
* Patients who are in private treatment
* Patients with high probability of loss to follow up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Life Quality | The change from basal point to 2, 6 and 12 months
  Change in the scale SF-36

SECONDARY OUTCOMES:
Use of pharmacotherapy and sanitary services | The change from baseline point to 12 months
  Change from basal point to one year in the use of pharmacotherapy and the use of sanitary services in primary care.

CONTACTS AND LOCATIONS:
Overall Officials: Amale Jauregui, Principal Investigator — Health Basdque Service
Locations (3):
- Spain (3):
  - Comarca Ezkerraldea, Barakaldo, Bizkaia
  - Comarca Bilbao, Bilbao, Bizkaia
  - Comarca Uribe, Leioa, Bizkaia

REFERENCES:
- [Derived] Jauregui A, Ponte J, Salgueiro M, Unanue S, Donaire C, Gomez MC, Burgos-Alonso N, Grandes G; Representing the PSICCAPAD Group. Efficacy of a cognitive and behavioural psychotherapy applied by primary care psychologists in patients with mixed anxiety-depressive disorder: a research protocol. BMC Fam Pract. 2015 Mar 20;16:39. doi: 10.1186/s12875-015-0248-3. PMID 25879932